CLINICAL TRIAL: NCT00210132
Title: Randomized Trial to Evaluate the Analgesic Efficacy of Inter Pleural Ropivacaine Road in Post Thoracotomy Pain for Oncologic Surgery
Brief Title: Analgesic Efficacy of Inter Pleural Ropivacaine Road in Post Thoracotomy Pain for Oncologic Surgery
Acronym: ROPAL-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IB2003-23
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Results first posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Pain; Cancer
Keywords: Thoracic surgery; postoperative pain; ropivacaine; inter pleural analgesia
MeSH Terms: conditions — Pain, Postoperative; Neoplasms | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Individual series of products were prepared by the Pharmacy according to a list (randomization list pre-established by the biostatistics department), which was not accessible to anyone until the results were analyzed. The treatments were sent by the pharmacy to the operating room in the form of pre-filled syringes with no distinguishing marks indicating the treatment group. Blindness was maintained during the evaluation period.

ARMS (2):
- Ropivacaine Arm (Experimental): ropivacaine at 7.5 mg/ml: 4 ml + 4 ml of saline solution to obtain 8 ml of a ropivacaine solution at 3.75 mg/ml injected into the intrapleural catheter every 6 hours.
  Treatment administration = every 6 hours for 48 hours.
  Interventions: Drug: Ropivacaine
- Reference Arm (Sham Comparator): 8 ml of saline solution will be injected into the intrapleural catheter. Treatment administration = every 6 hours for 48 hours.
  Interventions: Drug: Reference

INTERVENTIONS:
Drug: Ropivacaine — ropivacaine at 7.5 mg/ml: 4 ml + 4 ml of saline solution to obtain 8 ml of a ropivacaine solution at 3.75 mg/ml injected into the intrapleural catheter every 6 hours.
  Treatment administration = every 6 hours for 48 hours.
  Arms: Ropivacaine Arm
Drug: Reference — 8 ml of saline solution will be injected into the intrapleural catheter. Treatment administration = every 6 hours for 48 hours.
  Arms: Reference Arm

SUMMARY:
Thoracic surgery via posterolateral thoracotomy causes significant postoperative pain.

There are several methods of postoperative pain relief, including intravenous analgesics and local-regional analgesia techniques. Although thoracic epidural remains the gold standard, it is not without complications, which are rare but serious, and should be reserved for trained teams or patients with high morbidity.

Intrapleural analgesia is a simple method, performed by the surgeon intraoperatively.

Its effectiveness is controversial and the results remain inconsistent. Ropivacaine is a recently marketed local anesthetic with a modest vasoconstrictive effect. The variation in plasma levels of ropivacaine obtained by this technique has not yet been evaluated.

The purposes of this study are:

1. To determine the efficacy of inter pleural analgesia
2. To determine the plasmatic concentration of ropivacaine by inter pleural road

ELIGIBILITY:
Inclusion Criteria:

* Thoracotomy for oncology thoracic surgery
* Secondary or primary cancer
* American Society of Anesthesiology (ASA) class 1 or 2

Exclusion Criteria:

* Ropivacaine hypersensibility
* Psychiatric disorders
* Incapacity of using visual analog scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2003-10-01 (Actual); Primary Completion 2006-06-30 (Actual); Study Completion 2008-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre GEKIERE, MD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié - Centre Régional de Luttre Contre le Cancer de Bordeaux et du Sud Ouest, Bordeaux, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Ropivacaine Arm: ropivacaine at 7.5 mg/ml: 4 ml + 4 ml of saline solution to obtain 8 ml of a ropivacaine solution at 3.75 mg/ml injected into the intrapleural catheter every 6 hours.
  Treatment administration = every 6 hours for 48 hours.
  Ropivacaine: ropivacaine at 7.5 mg/ml: 4 ml + 4 ml of saline solution to obtain 8 ml of a ropivacaine solution at 3.75 mg/ml injected into the intrapleural catheter every 6 hours.
  Treatment administration = every 6 hours for 48 hours.
Period: Overall Study
Arm/Group | Ropivacaine Arm | Reference Arm
Started | 45 | 45
Completed | 44 | 41
Not Completed | 1 | 4
Not completed — Protocol Violation | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine Arm | Reference Arm | Total
Number analyzed (Participants) | 44 | 41 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (12.9) | 51.4 (13.6) | 53.9 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 11 | 30
  Male | 25 | 30 | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 44 | 41 | 85

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Major Post-operative Pain at Mobilization Following Lung Surgery by Posterolateral Thoracotomy
Description: Pain is measured using a visual analog scale (VAS), ranging from 0 (no pain) to 100 (worst pain ever).
  A participant is considered to have major pain if VAS score is >= 70.
Time Frame: Between surgery and up to 48 hours
Population: Participants with a VAS score available
Measure: Count of Participants; unit: Participants
Arm/Group | Ropivacaine Arm | Reference Arm
Number analyzed (Participants) | 41 | 39
Participants | 4 | 3
Statistical Analysis 1: Comparison: Ropivacaine Arm vs Reference Arm; Comparison of proportions; Test type: Superiority; p = 0.99, Fisher Exact

2. Secondary Outcome: Post-operative Morphine Consumption Following Lung Surgery by Posterolateral Thoracotomy
Description: Morphine consumption during the 48 hours following surgery. Morphine consumption is defined as the number of morphine boluses (1 bolus = 1mg).
Time Frame: between surgery and 48 hours
Population: Participants with available data at 48 hours.
Measure: Mean (Standard Deviation); unit: boluses
Arm/Group | Ropivacaine Arm | Reference Arm
Number analyzed (Participants) | 31 | 32
boluses | 29.9 (23.5) | 15.6 (17.4)
Statistical Analysis 1: Comparison: Ropivacaine Arm vs Reference Arm; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Ropivacaine Arm | Reference Arm
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/41
Other Adverse Events (participants affected / at risk) | 0/44 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes